CLINICAL TRIAL: NCT05871424
Title: Transdermal Buprenorphine Patch for Postoperative Pain Control in Laparoscopic Cholecystectomy: a Prospective Randomized, Placebo-controlled, Study
Brief Title: Transdermal Buprenorphine Patch for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3-2023-0007
Record Dates: First submitted 2023-03-12; First posted 2023-05-23 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buprenorphine patch group (Experimental)
  Interventions: Drug: buprenorphine patch group
- placebo group (Sham Comparator)
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: buprenorphine patch group — 5 mcg/h buprenorphine patch will be applied preoperatively
  Arms: buprenorphine patch group
Drug: placebo group — simple dressing tape only will be applied
  Arms: placebo group

SUMMARY:
Preliminary studies of the transdermal buprenorphine patch target chronic pain patients, and the pain relief effect and safety have been proven. There are previous reports that the transdermal buprenorphine patch is effective in acute postoperative pain control. However, no clinical studies have yet been reported on its application during laparoscopic cholecystectomy. Therefore, we designed this study to see if the use of a transdermal buprenorphine patch resulted in a better pain profile.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients 19 years of age or older who are expected to undergo laparoscopic cholecystectomy 2) ASA PS 1-3

Exclusion Criteria:

* (1) Patients with known hypersensitivity to buprenorphine, including patients with previous allergic contact dermatitis (2) Patients with drug resistance, opioid dependence, and treatment for drug withdrawal symptoms (3) Patients with severe respiratory dysfunction or respiratory depression (4) Patients currently taking other central nervous system depressants or muscle relaxants that may cause respiratory depression, hypotension, severe sedation, or lead to coma (5) If you are unable to read or understand the consent form (e.g. cognitive impairment, illiteracy, foreigners, etc.) (6) Other vulnerable subjects

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-06-11 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale pain score at movement | 6 hours after surgery
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Numeric rating scale pain score at rest | up to 2 weeks after the surgery
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) 1, 2, 6, 24, and 2 weeks after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No